CLINICAL TRIAL: NCT01163448
Title: Phase I Feasibility and Safety Study Using Preoperative High-Dose Single-Fraction Image-Guided Radiotherapy for Men Undergoing Radical Prostatectomy at High-Risk for Extraprostatic Cancer
Brief Title: Feasibility and Safety Study Using Preoperative High-Dose Single-Fraction Image-Guided Radiotherapy for Men Undergoing Radical Prostatectomy at High-Risk for Extraprostatic Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-013
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Prostate Cancer
Keywords: Prostate; Radiation; Radical prostatectomy; 09-013
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- High-Dose Single-Fraction Image-Guided Radiotherapy (Experimental): This will assess the feasibility and safety of this approach in men at high-risk for extraprostatic prostate cancer undergoing RP. This initial trial has been designed in a manner intended to emphasize patient comfort and safety.
  Interventions: Radiation: High-Dose Single-Fraction Image-Guided Radiotherapy for Men Undergoing Radical Prostatectomy

INTERVENTIONS:
Radiation: High-Dose Single-Fraction Image-Guided Radiotherapy for Men Undergoing Radical Prostatectomy — A baseline DCE-MRI will be obtained prior to the day of radiotherapy treatment. Immediately following the delivery of radiotherapy another DCE-MRI will be performed to assess for perfusion changes in the prostate resulting from irradiation. RP will be completed within 6 weeks (+ 2 weeks) of radiation and the RP specimen will be assessed for radiation treatment effect and other pathologic parameters (including surgical margin status) by a dedicated genitourinary pathologist. Following RP, participants will follow-up with their surgeon every 3 months for one year, with visits alternating between the urologist and the radiation oncologist. After the first year follow-up will occur at 6 month intervals until the patient is 3 years out from surgery.

SUMMARY:
This study is being done to test the safety of a single high-dose of radiation therapy before radical prostatectomy (removal of the prostate). The investigators want to find out what effects, good and/or bad, the radiation will have on men undergoing prostatectomy. The investigators are especially interested in men who are at risk for having cancer cells that have spread outside the prostate.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven prostate cancer verified at MSKCC. The biopsy will include a minimum of 10 cores
* Radical Prostatectomy (RP) chosen as the therapeutic method
* The size of the prostate will be < 70 cc by transrectal ultrasound or endorectal MRI imaging
* No radiographic evidence of lymph node metastases, bone metastases or soft tissue disease
* Risk of extraprostatic cancer of > 40% based on the MSKCC surgical nomogram
* Age > or = to 18 years
* KPS > or = to 80
* Able to tolerate immobilization cradle positioning

Exclusion Criteria:

* Allergic reaction to intravenous CT contrast (if premedicated, pt will not be excluded)
* Prior radiation to the planned target region
* Patients receiving concurrent chemotherapy
* Neoadjuvant hormonal therapy Luteinizing-hormone-releasing hormone(LHRH)agonist and/or antiandrogen)
* Prior transurethral resection of the prostate
* Normal tissue directly overlying target precluding ability to limit the bowel, bladder, rectum or other tissue to less than or equal to 15-16 Gy dose constraints
* Dominant prostatic lesion within 3 mm from the anterior rectal wall by imaging studies
* Creatinine clearance <60 ml/min/1.73m2

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility and safety of single-fraction image-guided intensity modulated radiotherapy (IG-IMRT). | 1 year
  Given prior to radical prostatectomy (RP) in men at high risk for extraprostatic cancer.

SECONDARY OUTCOMES:
To analyze the changes in prostate perfusion induced by single-fraction IG-IMRT. | 1 before radiation simulation, 1 after radiation treatment
  via dynamic contrast enhanced magnetic resonance imaging (DCE-MRI)
To assess the long-term toxicity of intensity modulated radiotherapy (IG-IMRT) | weeks 3, 6, 9, 12, 18, 24, 30, and 36 months after RP
  Given prior to radical prostatectomy (RP) with respect to urinary function, erectile function, and bowel function.
To assess the effect of IG-IMRT on the anticipated positive margin rate at the time of RP. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: James Eastham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm